CLINICAL TRIAL: NCT03089775
Title: A Randomized, Controlled Study to Evaluate the Effect of Topically Applied BBI-2000 (5%) on Allergic Responses in Subjects With Contact Hypersensitivity to Diphencyprone
Brief Title: Evaluation of Safety and Efficacy of BBI-2000 in Treating and Preventing Contact Dermatitis
Acronym: BBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresh Tracks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-2000-CL-101
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Contact Dermatitis
Keywords: Contact; Treatment; Prevention; BBI-2000; Dermatitis; Allergic
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BBI-2000 (Experimental): Cohort A
  Interventions: Drug: BBI-2000
- Vehicle (Placebo Comparator): Cohort A
  Interventions: Drug: Vehicle
- Multiple treatments (Other): Cohort B
  Interventions: Drug: BBI-2000; Drug: Vehicle; Other: Multiple treatments

INTERVENTIONS:
Drug: BBI-2000 — Experimental
  Arms: BBI-2000; Multiple treatments
Drug: Vehicle — Vehicle Comparator
  Arms: Multiple treatments; Vehicle
Other: Multiple treatments — BBI-2000, Vehicle, Clobetasol Propionate, No treatment
  Arms: Multiple treatments

SUMMARY:
This two cohort study (Cohort A and B) is being conducted to assess the safety and efficacy of BBI-2000 for the prevention (Cohort A) and treatment (Cohort B) of delayed type hypersensitivity reaction.

DETAILED DESCRIPTION:
This two cohort (Cohort A and B) single-center, randomized, controlled study is being conducted to evaluate the safety and efficacy of BBI-2000 for the prevention (Cohort A) and treatment (Cohort B) of delayed type hypersensitivity (DTH) reactions.

Subjects in Cohort A will initially receive either pre-treatment with BBI-2000 or vehicle, on an area on the back. Diphencyprone (DPCP) will then be administered, via Finn chamber, to the same area on the back. The treated area will then be assessed to determine if BBI-2000 was effective in preventing a contact hypersensitivity reaction.

Cohort B will first be sensitized with DPCP as in Cohort A. Indicated regions of the back will then be challenged to illicit a DTH reaction. Following the challenge, indicated regions on the subject's back will be treated with either (A) BBI-2000, (B) vehicle, (C) no topical application or (D) clobetasol propionate. The efficacy of BBI-2000 will be evaluated by monitoring response of the area of contact hypersensitivity reaction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 65 years inclusive at the time of consent, and either female of non-reproductive potential or male.
* Subjects must be healthy, normal volunteers per physical exam, laboratory and EKG assessments

Exclusion Criteria:

* History of contact dermatitis to medical adhesive bandages or glue.
* Medical history of dermatographism.
* Any medical condition causing immunosuppression.
* Prior treatment or therapies or history of sensitivity to any of the study products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Number of adverse events in each study group | 4 weeks
  Comparison of the number and severity of adverse event between study groups
Vital signs, physical examinations, ECG, blood analysis, urine analysis | 4 weeks
  Changes in vital signs, physical examinations, ECG, blood and urine analyses between study groups
Size of contact hypersensitivity reaction | 4 weeks
  Mean diameter (mm) of the contact hypersensitivity reaction induced by DPCP for subjects randomized to BBI-2000 (5%) as compared with vehicle

SECONDARY OUTCOMES:
Dermal thickness | 4 weeks
  Contact hypersensitivity reactions will be quantified using a high-frequency 20-Megahertz (MHz) ultrasound scanner
Diameter (mm) of the contact hypersensitivity area | 4 weeks
  Mean diameter (mm) of the contact hypersensitivity reaction induced by DPCP for areas randomized to BBI-2000, as compared with vehicle, no treatment, and clobetasol propionate over time

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Romel, MS, Study Director — Fresh Tracks Therapeutics, Inc.
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No